CLINICAL TRIAL: NCT01713842
Title: Phase II Open 24 Weeks Study to Evaluate Effect and Safety of Tocilizumab as the First Line Therapy in Subjects With Polymyalgia Rheumatica (PMR)
Brief Title: Tocilizumab Effect iN pOlymyalgia Rheumatica
Acronym: TENOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB 11-075 TENOR
Record Dates: First submitted 2012-09-17; First posted 2012-10-25 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-01

CONDITIONS: Polymyalgia Rheumatica
Keywords: Tocilizumab; Polymyalgia Rheumatica; Glucocorticotherapy; PMR-AS
MeSH Terms: conditions — Polymyalgia Rheumatica

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TCZ (Experimental): Tocilizumab at week 0, week 4 and week 8 8mg/kg at each perfusion
  Interventions: Drug: TCZ

INTERVENTIONS:
Drug: TCZ — Tocilizumab at week 0, 4 and 8.

SUMMARY:
Phase 1:

Patients are treated with infusions of Tocilizumab (TCZ) for 3 months. Clinical evaluation is performed using PMR-AS.

The PMR-AS is computed by summing the 5 variables after multiplying by 0.1 for weighting purposes: PMR-AS (activity scale = AS) = C reactive protein (CRP) (mg/dl) + patient scale (VASp) (0-10 scale) + physician scale (VASph) (0-10 scale) + morning stiffness(MST) [min]×0.1) + elevation of upper limbs (EUL) (0-3 scale).

At the end of the phase 1,the patients stop TCZ and entered in phase 2 at week 12.

Phase 2:

All the patients are included in the phase 2 and treated with glucocorticoid (GC)for 3 months. Two arms are possible according to the PMR-AS. Either the classical GC treatment (0.3mg/kg), either a low dose group of GC(0.15mg/kg) .

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 years and 75 years included
* PMR-AS > 10
* PMR according to the Chuang criteria
* Evolving since less than 12 months
* Without Horton disease
* Able to understand and accept the study
* Agree to sign the inform consent form
* Without GC, or at least during 1 month and stop since 7 days before the inclusion.
* Stable dose of Nonsteroidal anti-inflammatory since 4 weeks before the inclusion.
* Birth controlled during all the study and 6 months after

Exclusion Criteria:

* Disagree to participated
* Unable to understand the study
* Participation to an other study in the 3 months before the inclusion
* Treated by GC at 0.3mg/kg/d in the past 7 days
* Less than 50 years old or more than 75 years old
* Uncontrolled dyslipidemia, high blood pressure or cardiovascular disease
* Histories of important allergy
* Historically positive test or test positive at screening for HIV-1 antibody, hepatitis B surface antigen, or hepatitis C antibody.
* Abnormal screening blood test : leukocyte count less than 3.5 × 109 cells/L, neutrophil count less than 2 × 109 cells/L, hemoglobin level less than 85 g/L, platelet count less than 100 × 109 cells/L, or hepatic aminotransferase or alkaline phosphatase levels greater than 3 times the upper limit of normal
* Other inflammatory rheumatic disease or connective disease
* Clinical evidence of significant unstable or uncontrolled acute or chronic diseases not due to PMR (eg. Cardiovascular, pulmonary, hematologic, gastrointestinal, hepatic, renal, neurological, malignancy or infectious diseases)
* Current drug or alcohol abuse
* Patients treated with an immunosuppressive agents in the past 4 weeks
* Live/attenuated vaccine in the past 4 weeks
* Clinical symptoms of giant cell arteritis
* History of infection or infestation in the past 3 months
* Active tuberculosis
* Planned surgical procedure
* History of malignant neoplasm within the last 5 years, except for adequately treated cancer of the skin (basal or squamous cell)
* History or current tumoral hematological disease
* Severe allergic or anaphylactic reactions about one of the TCZ component
* Pregnant women during the study and six month after the end of the study
* Breast feeding mother
* Dysthyroidia
* Unstable treatment by statin in the past 3 months
* Parkinson disease
* Fibromyalgia
* Peripheric arthritis
* Articular chondrocalcinosis or hydorxyapatites rhumatisms

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-07; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Efficacy at W12 | 12 Weeks
  PMR-AS at week 12

SECONDARY OUTCOMES:
Safety and efficacy during the study | Week 2,4,8,12,16,20 and 24
  * To maintain low disease activity (PMR-AS) in the low corticosteroid dose group from W12 to W24
  * On the inflammatory changes (synovitis, myositis, tenosynovitis aund bursitis) between baseline, W2 and 12 visualize by ultrasonography, MRI and Tep-Scan.
  * On sparing corticosteroid, with the comparison of the cumulative corticosteroid dosage beetwen the two groups of patients in the phase 2, W12 to 24.
  * On the circulating serum cytokines and immunoregulators (IL-6, IL-1, BLyS/BAFF, IL-6 receptor, gp130) and B cells receptors and on the phenotype of circulating T- and B-cells between baseline and W4 and 12 On inflammatory parameters (CRP and ESR) between baseline and W 2,4,8,12,16,20 and 24
  * On the quality of life of patients between baseline and W 4,12,16, 20 and 24
  * To evaluate the side-effects in relation to the use of Tocilizumab treatment. [ Time Frame: After first, second and third treatment and during follow up ]

CONTACTS AND LOCATIONS:
Overall Officials: Valérie DEVAUCHELLE, Pr, Principal Investigator — CHRU de Brest
Locations (3):
- France (3):
  - CHR d'Orléans, Orléans, France
  - Brest University Hospital, Brest
  - Nantes University Hospital, Nantes

REFERENCES:
- [Derived] Carvajal Alegria G, Garrigues F, Bettacchioli E, Loeuille D, Saraux A, Cornec D, Devauchelle-Pensec V, Renaudineau Y. Tocilizumab controls bone turnover in early polymyalgia rheumatica. Joint Bone Spine. 2021 May;88(3):105117. doi: 10.1016/j.jbspin.2020.105117. Epub 2020 Dec 7. PMID 33301930
- [Derived] Laporte JP, Garrigues F, Huwart A, Jousse-Joulin S, Marhadour T, Guellec D, Cornec D, Devauchelle-Pensec V, Saraux A. Localized Myofascial Inflammation Revealed by Magnetic Resonance Imaging in Recent-onset Polymyalgia Rheumatica and Effect of Tocilizumab Therapy. J Rheumatol. 2019 Dec;46(12):1619-1626. doi: 10.3899/jrheum.180958. Epub 2019 Mar 15. PMID 30877202
- [Derived] Devauchelle-Pensec V, Berthelot JM, Cornec D, Renaudineau Y, Marhadour T, Jousse-Joulin S, Querellou S, Garrigues F, De Bandt M, Gouillou M, Saraux A. Efficacy of first-line tocilizumab therapy in early polymyalgia rheumatica: a prospective longitudinal study. Ann Rheum Dis. 2016 Aug;75(8):1506-10. doi: 10.1136/annrheumdis-2015-208742. Epub 2016 Feb 29. PMID 26929219